CLINICAL TRIAL: NCT04478227
Title: Single Arm Prospective Open Label Pilot Study Evaluating Short-Term Safety and Efficacy of Romiplostim in Children With Inherited and Acquired Disorders of Hematopoietic Failure
Brief Title: TPO-Mimetic Use in Children for Hematopoietic Failure
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Anjali Sharathkumar (Other)
Collaborators: Amgen (Industry)
Responsible Party: Sponsor-Investigator, Anjali Sharathkumar, Clinical Professor, University of Iowa
Organization: University of Iowa (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 202004776
Record Dates: First submitted 2020-07-10; First posted 2020-07-20 (Actual); Last update posted 2024-07-30 (Actual); Status verified 2024-07

CONDITIONS: Bone Marrow Failure Disorders; Aplastic Anemia; Thrombocytopenia; Refractory Cytopenia of Childhood; Myelodysplastic Syndrome(MDS)
MeSH Terms: conditions — Bone Marrow Failure Disorders; Anemia, Aplastic; Thrombocytopenia; Myelodysplastic Syndromes | interventions — romiplostim

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm A (Experimental): Arm A will include acquired bone marrow failure (BMF) disorders including aplastic anemia, refractory cytopenia of childhood/Myelodysplastic Syndrome(MDS) without monosomy 7 and 5q deletion abnormalities, toxin induced myelosuppression due to infection and inherited cytopenia with or without involvement of other cell lines who are transfusion dependent and or showing progression to bone marrow failure.
  Arm A: Start at 5 microgram/kg/dose per week along with standard of care and escalate with 2.5 microgram/kg/dose increments (per week at physician's discretion depending on the clinical and laboratory response) (Maximum: 20 microgram/kg/dose) based on response for at least 24 weeks or until hematopoietic response is seen, whichever comes first. If patient shows response, therapy will be continued for a total of 52 weeks.
  Interventions: Drug: Romiplostim
- Arm B (Experimental): Arm B will include children with chemo and or radiotherapy induced thrombocytopenia/cytopenia and children undergoing stem cell transplantation (SCT).
  Arm B: Starting dose 2 microgram/kg/dose per week with increments at 1 microgram/kg/dose (Maximum: 10 micrograms/kg/dose) depending on the laboratory response.
  Interventions: Drug: Romiplostim

INTERVENTIONS:
Drug: Romiplostim — Nplate is a thrombopoietin receptor agonist indicated for the treatment of thrombocytopenia in patients with chronic immune (idiopathic) thrombocytopenic purpura (ITP) who have had an insufficient response to corticosteroids, immunoglobulins, or splenectomy.
  Other Names: Nplate

SUMMARY:
This is an open label, prospective Pilot interventional study will investigate the safety and efficacy of Romiplostim, thrombopoietin (TPO) mimetic, in children (ages: 0 to 21 years) with broad scope of bone marrow failure disorders including acquired and inherited conditions as a first line of therapy along with standard of care.

DETAILED DESCRIPTION:
This investigator-initiated study will investigate the safety and efficacy of Romiplostim, thrombopoietin (TPO) mimetic, in children (ages: 0 to 21 years) with broad scope of bone marrow failure disorders (BMF) including acquired and inherited conditions as a first line of therapy along with standard of care.

Objectives: Primary objectives are to evaluate safety and preliminary efficacy of Romiplostim in children with BMF. Methods: This open label, prospective Pilot interventional study has two arms.

Arm A will include acquired bone marrow failure (BMF) disorders including aplastic anemia, refractory cytopenia of childhood without monosomy 7 and 5q deletion abnormalities, toxin induced myelosuppression due to infection and inherited cytopenia with or without involvement of other cell lines who are transfusion dependent and or showing progression to bone marrow failure. Arm B will include children with chemo and or radiotherapy induced thrombocytopenia/cytopenia and children undergoing stem cell transplantation (SCT). Children with cancer predisposition and other morbidities which are considered significant by the investigator will be excluded from the study.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 0 to ≤ 21 years
2. Child should be receiving ongoing care with pediatric hematology/oncology providers
3. Those enrolled in Arm A of the study should have a confirmed diagnosis of any of the following

   a. aplastic anemia i. Diagnosis of severe Aplastic anemia (newly diagnosed or refractory based on history of prior treatments) is established if Bone marrow cellularity <25% or and at least two of the following criteria are met:- (i) absolute neutrophil count less than 0.5 × 10^9/L, (ii) platelet count less than 20 × 10^9/L, and (iii) reticulocyte count less than 20 × 10^9/L ii. Moderate aplastic anemia is defined as bone marrow cellularity <50 percent and depression of at least two out of three blood counts below the normal values: criteria are met:- (i) absolute neutrophil count less than 1.2x10^9/m3, (ii) platelet count less than 70x10^9/L, and (iii) anemia with hemoglobin less than or equal to 8.5 g/dL and absolute reticulocyte count less than or equal to 60x10^9/L in transfusion-dependent patients but not fulfilling the criteria of severe aplastic anemia

   b. refractory cytopenia of childhood without monosomy 7 or 5q- and without an evidence of cytogenetic abnormality with predisposition to leukemia

   c. myelo-suppression contributing to severe pancytopenia (absolute neutrophil count <0.5 x 10^3/mm^3; platelet count less than 20 × 10^9/L, and reticulocyte count less than 20 × 10^9/L secondary to any other drug or infection

   d. diagnosis of inherited bone marrow failure without chromosomal fragility disorder
4. Those enrolled in Arm B of the study should have a confirmed diagnosis of any of the following:

   1. myelo-suppression specifically thrombocytopenia as defined by primary oncologist in children with solid tumors secondary to chemotherapy or radiation therapy contributing to delay in chemotherapy
   2. patient undergoing stem cell transplantation and experiencing persistent thrombocytopenia. This will include children not requiring platelet transfusions with a platelet count of <10 x 109/L, as well as those requiring platelet transfusions (transfusion dependent) for prevention of bleeding diathesis regardless of their platelet count at the time of recruitment (note: due to delayed engraftment these patients may have a higher platelet count because of platelet transfusion needs at the time of recruitment).
5. Adequate organ function within 7 days of enrollment defined as:

   1. Creatinine: ≤ 2.0 mg/dL
   2. Hepatic function:

      * For arm A, elevation of liver enzymes is acceptable for patients with hepatitis induced SAA as long as patient does not have history of chronic liver problem. If necessary, liver biopsy will be performed.
      * For Arm B, elevation of liver enzymes will be accepted as long as no chronic liver problem. Liver biopsy will be performed if necessary.
6. Females of childbearing potential agree to use effective contraception during the study period and for 4 months after completion of therapy
7. Must be able to provide written and voluntary informed consent.

Exclusion Criteria:

1. Gestational age < 32 weeks or Age > 21 years at the time of study enrolment
2. Preexisting condition with predisposition for thrombosis
3. Diagnosis of bone marrow failure syndrome with cancer predisposition including chromosomal fragility disorders (Fanconi anemia, Bloom syndrome, Ataxia Telangiectasia) and other conditions with known association towards cancer predisposition
4. Presence of complex karyotype or monosomy 7 or 5q- or other cytogenetic abnormality with known predisposition to cancer.
5. Diagnosis of MDS with excess blasts in transformation
6. Female subjects who are nursing or pregnant (positive serum or urine β-human chorionic gonadotropin [β-hCG] pregnancy test) at screening or pre-dose on Day 1.
7. Current alcohol or drug abuse.
8. Treatment with an investigational drug within 30 days or 5 half-lives (whichever is longer) preceding the first dose of study medication.
9. Active and uncontrolled infections (e.g. sepsis, hepatitis B, hepatitis C).
10. Chronic liver disease ie. Fibrosis or cirrhosis
11. Subjects infected with Human Immunodeficiency Virus (HIV).
12. Have a known immediate or delayed hypersensitivity reaction or idiosyncrasy to drugs chemically related to Romiplostim that contraindicates the subjects' participation
13. Known history of sensitivity or allergy to the active substance, to any of the excipients, or to any E. coli-derived product.
14. Moribund status or concurrent hepatic, renal, cardiac, neurologic, pulmonary, infectious, or metabolic disease of such severity that it would preclude the patient's ability to tolerate protocol therapy, or that death within 7-10 days is likely.
15. Subjects who have participated in any study using an investigational drug during the previous 30 days.
16. Non-English-speaking families who cannot speak or read English

Ages: 0 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 15 (Actual)
Dates: Start 2020-08-18 (Actual); Primary Completion 2024-01-18 (Actual); Study Completion 2024-01-18 (Actual)

PRIMARY OUTCOMES:
Occurrence of treatment-related adverse events (AEs) according to NCI CTCAE v5.0 | During treatment and through 90 days following discontinuation of treatment
  Categorize and quantify AEs per CTCAE version 5.0
To estimate preliminary efficacy of Romiplostim as measured by improvement in hematopoiesis | By 24 weeks of therapy
  Improvement in at least one of the cell blood lineages by 24 weeks of therapy:
  1. Platelet response (increase to 10 X 103/mL above baseline or stable platelet counts with transfusion independence for a minimum of 2 weeks in those who were transfusion dependent on entry into the protocol)
  2. Erythroid response (when pretreatment hemoglobin was, below 7 g/dL, defined as an increase in hemoglobin by 1.5 g/dL or, in transfused patients, a reduction in the units of packed red blood cell transfusions by an absolute number of at least 4 transfusions for 8 consecutive weeks, compared with the pretreatment transfusion number in the previous 8 weeks)
  3. Neutrophil response (when pretreatment absolute neutrophil count [ANC] of 0.5 x103 /mL as at least a 100% increase in ANC, or an ANC increase by 0.5 x103 /mL)

SECONDARY OUTCOMES:
To assess time to hematological response | Time from Romiplostim initiation to response, by 24 weeks of therapy
  Time from Romiplostim initiation to response, as defined in Outcome 2, for each cell lineage
To assess longitudinal changes in blood counts | From treatment beginning to end, up to 52 weeks
  Change in blood counts from Romiplostim initiation until the end of treatment
To assess the incidence of bleeding (including muco-cutaneous bleeding) | From treatment beginning to end, up to 52 weeks
  Occurrences of bleeding as defined by the International Society of Haemostasis and Thrombosis Bleeding Assessment Tool (https://bleedingscore.certe.nl/)
To assess the incidence of neutropenic fever | From treatment beginning to end, up to 52 weeks
  Number of occurrences of neutropenic fever
To assess the requirement of blood product support | Prior to initiation of treatment through end of treatment, up to 52 weeks
  Change in number of platelet and red call transfusions without active bleeding diathesis
To assess development of bone marrow myelofibrosis | at 3 to 6 months after treatment initiation; within 4 to 6 weeks after discontinuation of treatment or any other time-point if deemed clinically indicated
  Increase in bone marrow myelofibrosis as measured by reticulin staining of bone marrow biopsy at diagnosis and follow up bone marrow testing upon initiation of Romiplostim
To assess transfusion dependence or decreased platelet transfusion requirement among subjects who receive pretreatment platelet transfusion | Up to 24 weeks after treatment initiation
  Number of patients who are transfusion dependent or who require decreased platelet transfusion

CONTACTS AND LOCATIONS:
Overall Officials: Anjali A. Sharathkumar, MBBS, MD, MS, Principal Investigator — University of Iowa
Locations (1):
- University of Iowa Hospitals & Clinics, Iowa City, Iowa, United States

IPD SHARING:
Plan to Share IPD: No